CLINICAL TRIAL: NCT03402334
Title: Assessing Healthcare Outcomes of Hepatitis C Virus (HCV) Positive Patients Counseled for Cardiovascular Disease Risk Factors
Brief Title: Counseling Hepatitis C Virus (HCV) Positive Patients for Cardiovascular Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-610
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hepatitis C; Atherosclerosis
MeSH Terms: conditions — Hepatitis C; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: This is a two-arm study. Group A will receive the intervention in addition to standard of care counseling while Group B will receive only standard of care counseling.
Who Masked: Participant
Masking Description: Single-blinded study. Participants are blinded to their designation in the study arms. Investigators cannot be blinded since the intervention they are providing is patient counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVD risk factor counseling (Experimental): This arm will receive intervention 'Patient counseling for HCV associated CVD risk factors' in addition to standard of care Hepatitis C counseling.
  Cardiovascular risk factor counseling will include:
  1. Increased risk for atherosclerosis with chronic HCV infection
  2. Increased risk of heart attack and stroke
  3. Treatment of HCV infection and reduction of viral load reducing risk of stroke and heart attack
  Interventions: Behavioral: Patient counseling for HCV associated CVD risk factors
- Standard of care counseling (No Intervention): This arm will receive standard of care Hepatitis C counseling:
  1. HCV infection poses an increased risk for hepatocellular carcinoma
  2. Hepatitis C is a curable disease
  3. Hepatitis C is transmitted through blood to blood contact, primarily through sharing needles
  4. HCV+ individuals should be vaccinated for Hepatitis A (HAV) and Hepatitis B (HBV)
  5. HCV+ individuals should reduce alcohol intake and shellfish consumption

INTERVENTIONS:
Behavioral: Patient counseling for HCV associated CVD risk factors — Patients will be counseled for cardiovascular disease risk factors associated with Hepatitis C infection. Such risk factors include atherosclerosis, heart attack, and stroke. Cardiovascular risk factors can be managed through connection with primary care and reduced through curative HCV treatment.
  Arms: CVD risk factor counseling

SUMMARY:
The study aims to compare the effect of a cardiovascular education package intervention on treatment-seeking behavioral outcomes of HCV+ patients. This prospective multicenter trial will compare outcomes between the intervention group (HCV+ patients receiving the enhanced education package) and the control group (HCV+ patients receiving the standard of care, the basic education package). The primary outcome measured will be successful linkage to hepatology for a discussion of HCV treatment options. The secondary outcome measured will be linkage to primary care for chronic disease management.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD), including atherosclerosis, are now the leading causes of mortality both in the United States and globally. Unfortunately, the major risk factors that have been targeted by public health programs are all behavioral, and have not met with enough success. Hence, there is an acute need for more tangible interventions that afford new options to reduce disease burden from atherosclerosis.

While the association of Hepatitis C virus (HCV) infection with life threatening complications such as liver cirrhosis and hepatocellular carcinoma (HCC) is well established, the recent discovery of HCV as a risk factor for atherosclerosis presents a new target for CVD control. In the largest epidemiological study of HCV and cardiovascular disease to date, HCV positive individuals were determined to have a significantly higher incidence of myocardial infarction, congestive heart failure, and corrective procedures for coronary artery disease including bypass grafting and angioplasty (1). Subsequent meta- analyses have lent increasing support to this relationship, showing adjusted odds ratios (OR) of 1.76 - 2.24 of carotid atherosclerosis in HCV+ patients (2,3).

The epidemiological evidence supporting the link of HCV and atherosclerosis has been further supported by bench research elucidating the role of HCV in vascular cytotoxicity and systemic inflammation. HCV viral replication has been shown within carotid artery plaques (4), as a result of viral endocytosis through the LDL receptor (5). HCV promotes intracellular oxidative stress, monocyte recruitment, and subsequent endothelial dysfunction leading to the promotion of atherosclerosis (6). In addition, HCV infection leads to a systemic inflammatory state promoting the acceleration of arterial vascular disease (7,8). Robust evidence now supports HCV as strongly pro-atherogenic (2,9), a relationship that is irrespective of HCV genotype or degree of histological liver pathology (10).

Viral RNA load of Hepatitis C has been shown to directly correlate with the atherosclerotic burden (10,11). HCV RNA levels are associated with advanced phase carotid plaques and carotid intima-media thickness (10). In addition, HCV RNA has been found in direct association with serum fibrinogen and C-reactive protein levels, which in turn were independently associated with carotid atherosclerosis (10). Together, such data suggest that managing HCV viral load will, in turn, control the cardiovascular manifestations of this disease.

Similar to atherosclerotic burden, higher viral loads correlate well with increased risk of cardiovascular and cerebrovascular associated mortality (2,9,11). Recent meta-analyses show the HCV+ population with an adjusted OR of 1.3 to 1.97 for cerebrovascular incidents (12) and an adjusted OR of 1.65 for death due to cardiovascular disease (3). Of importance, combination ribavirin and interferon therapy has been shown to decrease such non-hepatic mortality as well as incidence of stroke in HCV+ patients (13,14). Thus, prompt and effective management of HCV can lead to suppression of viral loads, which can result in decreased mortality secondary to cardiovascular events (9,10).

Current estimates indicate that 3.2 million people living in the United States are HCV-infected, a disease that has now surpassed HIV in annual mortality (15,16). The development of combination sofosbuvir and ledipasvir (Harvoni), a direct acting, non-interferon based therapy, has made HCV a newly curable disease. This is an exciting new field with potential for a novel anti-viral intervention to reduce the burden of atherosclerosis and the associated deaths from ischemic heart disease and strokes.

Goal: To investigate the role of HCV treatment in decreasing atherosclerotic co-morbidities.

Specific Aim 1 For HCV: To increase HCV healthcare-seeking behavior of HCV+ patients by educating them about their increased risk for atherosclerosis, cardiovascular disease, and cerebrovascular events.

Specific Aim 2 For Atherosclerosis: To positively influence HCV+ patients to follow up with a primary care physician for either prevention or management of any potential atherosclerotic comorbidities.

Methodology Tulane Medical students trained by the New Orleans Office of Public Health (OPH) currently provide HCV screening and counseling across six New Orleans community health clinics: Ozanam Inn, New Orleans Mission, Bethel Colony South, Grace House, St. Anna's Mobile Clinic, and Ruth Fertel. HCV+ patients are linked to a primary care physician (PCP) at Healthcare for the Homeless (HCH), and in addition, curative HCV treatment at University Medical Center (UMC) Hepatology Clinic. Since its inception in 2015, 936 patients have been tested through this rapidly growing community program.

A randomized controlled trial will be conducted. The control will receive the current standard of care in those clinics, including the "basic education package" on HCV-associated cirrhosis and HCC. The intervention group will receive an "augmented education package" that includes all the components of the basic package, plus education on atherosclerosis and associated cardiovascular risk. All HCV + patients will be referred to a single PCP for screening, prevention, or management of atherosclerosis. Statistical data analysis will be done using Statistical Analysis Software.

For Study Aim 1 Outcome Measures for HCV: The percentage of patients attending their subsequent UMC hepatology appointment for the treatment and control groups will be measured, indicating the effectiveness of the "augmented education package" at improving patients' willingness to treat their HCV infection.

For Study Aim 2 Outcome Measures for Atherosclerosis: Patients referred to the PCP will be tracked to assess the proportion that attended their PCP appointment, measuring the impact of the "augmented education package" at positively influencing HCV+ patients to follow up with primary care for their atherosclerotic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* HCV antibody positive tested at one of six locations in New Orleans: Ozanam Inn, New Orleans Mission, Bethel Colony South, Grace House, St. Anna's Mobile Clinic, and Ruth Fertel

Exclusion Criteria:

* vulnerable populations including children, prisoners, pregnant women
* non-English speaking patients since effective counseling cannot be provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Linkage to HCV Care | Patient will be assessed for follow up within 6 months post counseling
  The percentage of patients attending their subsequent University Medical Center hepatology appointment for the treatment and control groups will be measured, indicating the effectiveness of the "augmented education package" at improving patients' willingness to treat their HCV infection.

SECONDARY OUTCOMES:
Linkage to Primary Care | Patient will be assessed for follow up within 6 months post counseling
  Patients referred to the primary care provider (PCP) will be tracked to assess the proportion that attended their PCP appointment, measuring the impact of the "augmented education package" at positively influencing HCV+ patients to follow up with primary care for their atherosclerotic comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Austin T Jones, MD, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University HCV Testing Clinics, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be disclosed

REFERENCES:
- [Background] Butt AA, Xiaoqiang W, Budoff M, Leaf D, Kuller LH, Justice AC. Hepatitis C virus infection and the risk of coronary disease. Clin Infect Dis. 2009 Jul 15;49(2):225-32. doi: 10.1086/599371. PMID 19508169
- [Background] Huang H, Kang R, Zhao Z. Is hepatitis C associated with atherosclerotic burden? A systematic review and meta-analysis. PLoS One. 2014 Sep 3;9(9):e106376. doi: 10.1371/journal.pone.0106376. eCollection 2014. PMID 25184517
- [Background] Petta S, Maida M, Macaluso FS, Barbara M, Licata A, Craxi A, Camma C. Hepatitis C Virus Infection Is Associated With Increased Cardiovascular Mortality: A Meta-Analysis of Observational Studies. Gastroenterology. 2016 Jan;150(1):145-155.e4; quiz e15-6. doi: 10.1053/j.gastro.2015.09.007. Epub 2015 Sep 18. PMID 26386298
- [Background] Boddi M, Abbate R, Chellini B, Giusti B, Giannini C, Pratesi G, Rossi L, Pratesi C, Gensini GF, Paperetti L, Zignego AL. Hepatitis C virus RNA localization in human carotid plaques. J Clin Virol. 2010 Jan;47(1):72-5. doi: 10.1016/j.jcv.2009.10.005. Epub 2009 Nov 5. PMID 19896417
- [Background] Germi R, Crance JM, Garin D, Guimet J, Lortat-Jacob H, Ruigrok RW, Zarski JP, Drouet E. Cellular glycosaminoglycans and low density lipoprotein receptor are involved in hepatitis C virus adsorption. J Med Virol. 2002 Oct;68(2):206-15. doi: 10.1002/jmv.10196. PMID 12210409
- [Background] Cuciureanu T, Chiriac S, Chiorescu M, Girleanu I, Trifan A. Chronic hepatitis C virus infection: a new modifiable cardio-metabolic risk factor? Clujul Med. 2017;90(3):251-255. doi: 10.15386/cjmed-793. Epub 2017 Jul 15. PMID 28781519
- [Background] Adinolfi LE, Zampino R, Restivo L, Lonardo A, Guerrera B, Marrone A, Nascimbeni F, Florio A, Loria P. Chronic hepatitis C virus infection and atherosclerosis: clinical impact and mechanisms. World J Gastroenterol. 2014 Apr 7;20(13):3410-7. doi: 10.3748/wjg.v20.i13.3410. PMID 24707124
- [Background] Munoz M, Liesenfeld O, Heimesaat MM. Immunology of Toxoplasma gondii. Immunol Rev. 2011 Mar;240(1):269-85. doi: 10.1111/j.1600-065X.2010.00992.x. PMID 21349099
- [Background] Voulgaris T, Sevastianos VA. Atherosclerosis as Extrahepatic Manifestation of Chronic Infection with Hepatitis C Virus. Hepat Res Treat. 2016;2016:7629318. doi: 10.1155/2016/7629318. Epub 2016 Jan 13. PMID 26885388
- [Background] Adinolfi LE, Restivo L, Zampino R, Guerrera B, Lonardo A, Ruggiero L, Riello F, Loria P, Florio A. Chronic HCV infection is a risk of atherosclerosis. Role of HCV and HCV-related steatosis. Atherosclerosis. 2012 Apr;221(2):496-502. doi: 10.1016/j.atherosclerosis.2012.01.051. Epub 2012 Feb 8. PMID 22385985
- [Background] Lee MH, Yang HI, Wang CH, Jen CL, Yeh SH, Liu CJ, You SL, Chen WJ, Chen CJ. Hepatitis C virus infection and increased risk of cerebrovascular disease. Stroke. 2010 Dec;41(12):2894-900. doi: 10.1161/STROKEAHA.110.598136. Epub 2010 Oct 21. PMID 20966408
- [Background] He Huang, Kang R, Zhao Z. Hepatitis C virus infection and risk of stroke: a systematic review and meta-analysis. PLoS One. 2013 Nov 12;8(11):e81305. doi: 10.1371/journal.pone.0081305. eCollection 2013. PMID 24265844
- [Background] Hsu CS, Kao JH, Chao YC, Lin HH, Fan YC, Huang CJ, Tsai PS. Interferon-based therapy reduces risk of stroke in chronic hepatitis C patients: a population-based cohort study in Taiwan. Aliment Pharmacol Ther. 2013 Aug;38(4):415-23. doi: 10.1111/apt.12391. Epub 2013 Jun 26. PMID 23802888
- [Background] Berenguer J, Rodriguez E, Miralles P, Von Wichmann MA, Lopez-Aldeguer J, Mallolas J, Galindo MJ, Van Den Eynde E, Tellez MJ, Quereda C, Jou A, Sanz J, Barros C, Santos I, Pulido F, Guardiola JM, Ortega E, Rubio R, Jusdado JJ, Montes ML, Gaspar G, Esteban H, Bellon JM, Gonzalez-Garcia J; GESIDA HIV/HCV Cohort Study Group. Sustained virological response to interferon plus ribavirin reduces non-liver-related mortality in patients coinfected with HIV and Hepatitis C virus. Clin Infect Dis. 2012 Sep;55(5):728-36. doi: 10.1093/cid/cis500. Epub 2012 May 18. PMID 22610932
- [Background] Klevens RM, Hu DJ, Jiles R, Holmberg SD. Evolving epidemiology of hepatitis C virus in the United States. Clin Infect Dis. 2012 Jul;55 Suppl 1(Suppl 1):S3-9. doi: 10.1093/cid/cis393. PMID 22715211
- [Background] Ly KN, Xing J, Klevens RM, Jiles RB, Ward JW, Holmberg SD. The increasing burden of mortality from viral hepatitis in the United States between 1999 and 2007. Ann Intern Med. 2012 Feb 21;156(4):271-8. doi: 10.7326/0003-4819-156-4-201202210-00004. PMID 22351712